CLINICAL TRIAL: NCT05880108
Title: Modifying Adiposity Through Behavioral Strategies to Improve COVID-19 Rehabilitation
Acronym: MARVEL
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Collaborators: Baltimore VA Medical Center (U.S. Federal Agency); South Texas Veterans Health Care System (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: F4572-R; 1I01RX004572-01A1 (NIH)
Record Dates: First submitted 2023-05-25; First posted 2023-05-30 (Actual); Last update posted 2025-06-29 (Actual); Status verified 2025-06

CONDITIONS: Post-COVID Conditions; Obesity
Keywords: COVID-19; Obesity; Senescence; Weight Loss; Exercise
MeSH Terms: conditions — Post-Acute COVID-19 Syndrome; Obesity; COVID-19; Weight Loss; Motor Activity

STUDY DESIGN:
Intervention Model Description: Weight Loss Program (Diet and Exercise)
Who Masked: Outcomes Assessor
Masking Description: Outcome assessors will be blinded to treatment allocation/group assignment
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Weight Loss (Experimental): Participants will be asked to participate in a 1x/week center-based or tele-health nutrition diet class, 2x/week center-based exercise classes, and 1x/week exercise session conducted on their own for approximately 12 weeks.
  Interventions: Behavioral: 12-weeks of Weight Loss
- Weight Stability (Active Comparator): Participants will be asked to participate in a 1x/week center-based or tele-health education class, 2x/week center-based or tele-health stretching/balance classes, and 1x/week stretching/balance session conducted on their own for approximately 12 weeks.
  Interventions: Behavioral: 12-weeks of Weight Stability

INTERVENTIONS:
Behavioral: 12-weeks of Weight Loss — Participants will be asked to participate in a 1x/week center-based or tele-health nutrition diet class, 2x/week center-based exercise classes, and 1x/week exercise session conducted on their own for ~12 weeks.
  Arms: Weight Loss
Behavioral: 12-weeks of Weight Stability — Participants will be asked to participate in a 1x/week center-based or tele-health education class, 2x/week center-based stretching/balance classes, and 1x/week stretching/balance session conducted on their own for ~12 weeks.
  Arms: Weight Stability

SUMMARY:
The research in this VA Merit will examine the effects of obesity and Post-COVID Conditions (PCC) on physical functioning, health-related quality of life, and adipose tissue inflammatory and cellular senescence profiles in older Veterans. Further, it will evaluate whether a weight loss intervention, including dietary modification and exercise, in obese Veterans with and without PCC will reduce systemic and adipose tissue inflammation and senescence and promote PCC recovery.

DETAILED DESCRIPTION:
Findings of post-acute sequelae of Post-COVID Conditions (PCC) manifestations of fatigue, pain, dyspnea, and muscle weakness, provide a strong rationale for rehabilitation; yet few formal studies exist and the effects of severe acute respiratory syndrome coronavirus-2 infection on function are not well described. Notably, two-thirds of Veterans are overweight and obese, rendering excess adiposity a significant risk factor and a high-priority area related to PCC prevention and care. Obesity increases the risk of severe illness in Veterans recovering from PCC, but how it does so is not fully understood.

Recent research suggests that excess adipose tissue is associated with adverse changes in adipose cellular function, and that these variations may be involved in the biology of aging and the etiology of aging-related diseases. Adipose tissue contains cells that have undergone cellular senescence, which induces inflammation, cytotoxicity, and metabolic dysfunction in other cells and tissues. However, the precise role of adipose tissue cellular composition on PCC recovery is limited.

Thus, the investigators propose to evaluate the role of obesity and PCC on physical functioning, health-related quality of life (HRQOL), and systemic and adipose tissue inflammatory and cellular senescence profiles in ethnically diverse older Veterans from the Audie Murphy (San Antonio) and Baltimore VA Medical Centers. Further, the investigators propose a randomized controlled trial to determine whether a reduction in body weight and increased physical function by a weight loss intervention (WL), including dietary modification and exercise, in obese Veterans with PCC will reduce systemic and adipose tissue inflammation and senescence, which will have important implications for PCC recovery.

ELIGIBILITY:
Inclusion Criteria:

1. U.S. Veteran
2. Self-reported COVID-19 naïve or COVID-19 > 90 days ago for lean and obese PCC naïve or documented COVID-19 for the lean and obese PCC groups (At least one PCC symptom >4 weeks)
3. Body Mass Index: 19-25 or 30-50 kg/m2

Exclusion Criteria:

1. Neurologic, musculoskeletal, or other condition that limits subject's ability to complete study physical assessments
2. Active inflammatory, COVID-19, autoimmune, infectious, hepatic (LFTs > 2.5 x WNL), renal (eGFR<45), gastrointestinal, malignant, and psychiatric disease
3. Uncontrolled diabetes (HbA1c >10% or the current use of insulin)
4. Weight change within the past month of >5 kg
5. Self-reported alcohol or drug abuse
6. Anti-coagulant medication usage

Max Age: 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2024-06-03 (Actual); Primary Completion 2028-09-30 (Estimated); Study Completion 2028-09-30 (Estimated)

PRIMARY OUTCOMES:
Cardiorespiratory Fitness (VO2max) | Baseline
  VO2max (ml/kg/min) comparison between lean PCC naïve, lean with PCC, obese PCC naïve, and obese with PCC

SECONDARY OUTCOMES:
Change in Cardiorespiratory Fitness (VO2max) | Baseline, After 12 weeks of Weight Loss
  Change in VO2max (L/min)
Change in adipose tissue cellular senescence | Baseline, After 12 weeks of Weight Loss
  Change in adipose tissue chemokine (C-C motif) ligand 3 (CCL3)

CONTACTS AND LOCATIONS:
Overall Officials: Alice S. Ryan, PhD, Principal Investigator — Baltimore VA Medical Center VA Maryland Health Care System, Baltimore, MD
Locations (2):
- United States (2):
  - Baltimore VA Medical Center VA Maryland Health Care System, Baltimore, MD, Baltimore, Maryland
  - South Texas Health Care System, San Antonio, TX, San Antonio, Texas

IPD SHARING:
Plan to Share IPD: No